CLINICAL TRIAL: NCT03061656
Title: High-dose 131I-MIBG Treatment Incorporated Into Tandem High-dose Chemotherapy and Autologous Stem Cell Transplantation in Patients With High-risk Neuroblastoma
Brief Title: Tandem High Dose Chemotherapy With 131I-MIBG Treatment in High Risk Neuroblastoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Ministry of Health, Republic of Korea (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-10-020
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: High Risk Neuroblastoma
MeSH Terms: interventions — Cyclophosphamide; Carboplatin; Etoposide; 3-Iodobenzylguanidine; Thiotepa; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High risk neuroblastoma (Experimental): 1. Conventional chemotherapy (9 cycles)
  2. Surgery conventional chemotherapy (after 6 cycles of chemotherapy)
  3. Tandem HDCT/autoSCT
     * First HDCT (cyclophosphamide, etoposide, carboplatin)
     * Second HDCT (high-dose 131I-MIBG, thiotepa, melphalan)
  4. Local radiotherapy
  5. Retinoic acid, interleukin-2
  Interventions: Drug: Cyclophosphamide; Drug: Carboplatin; Drug: Etoposide; Radiation: 131I-MIBG; Drug: Thiotepa; Drug: Melphalan

INTERVENTIONS:
Drug: Cyclophosphamide — 1st HDCT
Drug: Carboplatin — 1st HDCT
Drug: Etoposide — 1st HDCT
Radiation: 131I-MIBG — 2nd HDCT
Drug: Thiotepa — 2nd HDCT
Drug: Melphalan — 2nd HDCT

SUMMARY:
The purpose of this study is to evaluate the efficacy and toxicity of tandem HDCT/ASCT including high-dose 131I-metaiodobenzylguanidine (MIBG) treatment. In the present study, a single arm trial of tandem HDCT/ASCT will be carried out.

DETAILED DESCRIPTION:
Although the outcome of high-risk neuroblastoma has improved after the introduction of HDCT/ASCT, the outcome was still unsatisfactory with 30-40% of survival. We previously reported the results of a single arm prospective trial (SMC NB-2004 study) using tandem HDCT/auto-SCT for high-risk neuroblastoma. In the NB-2004 trial, total body irradiation (TBI) was incorporated in second transplantation. Survival rates were very encouraging; however, short- and long-term toxicities associated with tandem HDCT/auto-SCT, particularly TBI, were also very significant. For this reason, we designed a new prospective trial (SMC NB-2009 study), in which only TBI in the second HDCT/auto-SCT of NB-2004 study was substituted with high-dose 131I-MIBG treatment in order to reduce short- and long-term toxicities without jeopardizing survival rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high-risk neuroblastoma

Exclusion Criteria:

* Patients with progressive disease before high-dose chemotherapy
* Patients whose parents want to stop or change the planned treatment
* Patients with organ toxicities of NCI grade >2 before high-dose chemotherapy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of event free survival | Up to 5 years
  Event is defined as relapse, disease progression or treatment-related mortality.

SECONDARY OUTCOMES:
Rate of treatment-related adverse events as assessed by CTCAE v4.0 | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ki Woong Sung, Principal Investigator — Samsung Medical Center

REFERENCES:
- [Derived] Lee JW, Lee S, Cho HW, Ma Y, Yoo KH, Sung KW, Koo HH, Cho EJ, Lee SK, Lim DH. Incorporation of high-dose 131I-metaiodobenzylguanidine treatment into tandem high-dose chemotherapy and autologous stem cell transplantation for high-risk neuroblastoma: results of the SMC NB-2009 study. J Hematol Oncol. 2017 May 16;10(1):108. doi: 10.1186/s13045-017-0477-0. PMID 28511709